CLINICAL TRIAL: NCT01481142
Title: Multicentre Investigation of the Efficacy and Safety of Adacolumn® GMA in Patients With Steroid-Dependent Active Ulcerative Colitis and Insufficient Response or Intolerance to Immunosuppressants and/or Biological Therapies
Brief Title: Adacolumn in Refractory UC Patients Trial
Acronym: ART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ada-UC-08-102
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Ulcerative Colitis, Active Moderate
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adacolumn (Experimental)
  Interventions: Device: (GMA) Adsorptive Apheresis

INTERVENTIONS:
Device: (GMA) Adsorptive Apheresis — Patients will be treated with once-weekly Adacolumn® apheresis over 5 consecutive weeks; treatment can be extended to up to 10 treatments administered once weekly over 10 weeks.

SUMMARY:
The objectives of the study are to observe and document the efficacy and safety of 5 or more Adacolumn treatments, administered once weekly over 5 or more weeks, in a specific subset of ulcerative colitis patients. The patient subset of interest is those with moderate/severe, steroid-dependent, active ulcerative colitis with insufficient response or intolerance to immunosuppressants and/or biological agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled into the study will be between 18 and 75 years old and have moderate to severe, steroid-dependent, active ulcerative colitis documented by clinical symptoms, endoscopic findings and histology. Patients will have an ulcerative colitis clinical activity (CAI) of ≥6 and an endoscopic activity index (EAI) of ≥4. Patients will have an insufficient response or intolerance to immunosuppressants and/or biological treatment agents. Patients are required to have adequate peripheral venous access to allow completion of apheresis treatment.

Exclusion Criteria:

- A patient will be excluded from the study if he/she meets any of the following criteria:

1. Is febrile (body temperature >38ºC).
2. Has evidence of toxic megacolon.
3. Has known obstructive disease of the gastrointestinal system.
4. Is anticipated to need surgery within the next 24 weeks.
5. Has a history of hypersensitivity reaction associated with an apheresis procedure or an intolerance to apheresis procedures.
6. Has proctocolectomy, total colectomy, ileostomy, stoma or ileal pouch-anal anastomosis.
7. Has a history of allergic reaction to heparin or of heparin-induced thrombocytopenia.
8. Has a known infection with enteric pathogens, pathogenic ova or parasites, or a positive test for cytomegalovirus.
9. Has symptomatic hypotension.
10. Has a history of physical findings consistent with a cerebrovascular accident.
11. Has a history of myocardial infarction or unstable angina within the previous 6 months.
12. Has undergone coronary artery bypass graft surgery or angioplasty within the previous 6 months.
13. Has congestive heart failure (New York Heart Association Class III or IV).
14. Has a prosthetic heart valve, pacemaker or other permanent implant.
15. Has severe cardiovascular or peripheral vascular disease.
16. Has liver disease defined as levels of aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) or alkaline phosphatase of greater than 2.5 × the upper limit of the normal range for the laboratory performing the test.
17. Has a history of cirrhosis.
18. Has a known bleeding disorder (prothrombin time [PT] or partial thromboplastin time [PTT] greater than 1.5 × the upper limit of the normal range for the laboratory performing the test) or requires concomitant anticoagulant therapy for purposes other than apheresis treatment.
19. Has a prior history suggestive of a hypercoagulable disorder, including 1 or more episodes of pulmonary embolism or deep vein thrombosis.
20. Has a known infection with hepatitis B or C or human immunodeficiency virus.
21. Has abnormal haematology parameters defined as severe anaemia with haemoglobin <8.5 g/dL, white blood cell count <3500/µL or granulocyte count <2000/µL.
22. Has a fibrinogen level >700 mg/dL.
23. Has renal insufficiency, defined as a serum creatinine level greater than 150% of the upper limit of the normal range for the laboratory performing the test.
24. Has had major surgery within the previous 6 weeks.
25. Has any of the following types of infection:

    * An active infection within 4 weeks of successful completion of antibiotic treatment for a bacterial infection.
    * Febrile viral infection within the 4 weeks prior to entry into the study.
    * Systemic fungal infection that required therapy which was completed within the 12 weeks prior to entry into the study.
26. Current drug or alcohol abuse.
27. Is pregnant, lactating or planning to become pregnant during the study.
28. Has used an investigational medicinal product, biologic agent or device within the last 30 days.
29. Adults lacking capacity who are unable to give consent by themselves due to physical and or mental incapacity.
30. Prisoners and patients who have undergone psychiatric treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the ulcerative colitis remission rate at Week 12, defined as a CAI (Rachmilewitz) score of ≤4. | 12 weeks

SECONDARY OUTCOMES:
Ulcerative colitis response rate at Week 12, with response defined as a reduction in CAI of ≥3. | 12 weeks
Response and remission rates at Weeks 24 and 48 | 12 weeks
Change from Baseline in CAI at Weeks 12, 24 and 48 | 12 weeks, 24 weeks and 48 weeks
Change from Baseline in EAI at Week 12 | 12 weeks
Time to remission and response | Baseline
The proportion of patients reaching steroid-free remission/steroid-free response at any visit and by visit at Weeks 12, 24 and 48. | 12 weeks, 24 weeks and 48 weeks
Time to steroid-free remission and response. | Baseline
Colectomy rate at Week 96 | 96 weeks
Change from Baseline in concomitant medication (steroid) dose at Weeks 12, 24 and 48. | 12 weeks, 24 weeks and 48 weeks
Quality of life changes based on the Short Health Scale for ulcerative colitis at Weeks 5, 12, 24 and 48. | 5 weeks, 12 weeks, 24 weeks and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Axel Dignass, Professor, Principal Investigator — Markus Krankenhaus
Locations (1):
- Clinique Universitaire d'Hépato-Gastroentérologie, Grenoble, France